CLINICAL TRIAL: NCT05453643
Title: EEG Analysis for the Objective Assessment of Secondary Hypersomnolence in Order to Limit the Accidental Risk
Brief Title: EEG Analysis for the Objective Assessment of Drowsiness
Acronym: MEEGASAFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Physip S.A (Industry)
Collaborators: University of Bordeaux (Other); National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MGSF
Record Dates: First submitted 2022-06-14; First posted 2022-07-12 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-07

CONDITIONS: Sleep Deprivation
Keywords: Sleep deprivation; Secondary hypersomnolence; Objective Sleepiness; Subjective Sleepiness; Cognitive performance; Driving
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep deprivation (Experimental): healthy volunteers
  Interventions: Behavioral: sleep deprivation patterns

INTERVENTIONS:
Behavioral: sleep deprivation patterns — Sleep deprivation patterns 1 (SDP1) ; total sleep deprivation for 24 hours followed by early morning sleep and an extended 17 hours wakefulness. Sleep deprivation patterns 2 (SDP2) : Sleep interrupted by two half-hour awakenings

SUMMARY:
The objective of this clinical study is to develop solutions for the evaluation and management of drowsiness, based on 2 EEG sensors only, aiming at reducing the risk of accidents related to secondary hypersomnolence (sleepiness induced by sleep restriction or abnormal sleep/wake cycle). This project will allow a better understanding of the determinants of drowsiness and its impact on cognitive performance and the development of methods and models for the evaluation and prediction of cognitive performance deficit related to sleepiness. The secondary hypersomnolence will be objectified by continuous EEG recording and analysed by visual reading according to Objective Sleepiness Scale (OSS) criteria and automatically analyzed using the MEEGAWAKE algorithm (developed by PHYSIP). The level of secondary hypersomnolence will be modified by varying the duration and maintening of prior sleep or the sleep timing. The ability to stay awake will be measured by the maintenance of wakefulness test (MWT). Subjective sleepiness and mind wandering will be measured before and/or after all measurements. Simulated driving task, maintenance of wakefulness tests and several cognitive tasks to measure sustained attention, alertness, selective attention will be performed every 4 hours.

DETAILED DESCRIPTION:
Chronotype and general tendency to daydream in daily life will be evaluated at the inclusion visit. Healthy volunteers will be placed in sleep deprivation patterns that will modify the level of secondary hypersomnolence. These patterns correspond to sleep deprivation caused by work schedules usually observed: shift work (SDP1) or night on-call (SDP2). shift work will be simulated by total sleep deprivation for 24 hours (comparable to the first day of a night worker) followed by early morning sleep, and an extended 17 hours wakefulness (comparable to second day of night shift). Secondary hypersomnolence will be assessed throughout prolonged awakenings (24 hours + 17 hours). The night on-call will be simulated by two half-hour awakenings during the nocturnal sleep. Hypersomnolence will be measured within 17 hours of wakefulness following this sleep fragmentation. The sleep history (quantity and quality of sleep) will be evaluated by actigraphy + ambulatory polysomnography (1 day before the experiment) and 2 polysomnographies in the laboratory during the experiment. Polysomnography recordings will be visually and automatically analyzed by the ASEEGA algorithm. Ambulatory recordings are automatically analyzed by ASEEGA. Throughout these sleep deprivation patterns, electrophysiological variables (EEG, EOG and EMG) will be continuously recorded in order to identify objective drowsiness states determined visually using the OSS or automatically by the MEEGAWAKE algorithm. Subjective sleepiness scale, Mind wandering scale, maintenance of wakefulness tests (MWT, electrophysiological test) and cognitive tests will be repeated, every 4hr, throughout the sleep deprivation patterns in order to determine abilities to stay awake, driving performance, sustained and selective attention, vigilance.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 27,
* With a score on the PHQ-4 scale less than or equal to 2 for scores A (Anxiety) and D (Depression),
* Subjects with no complaints of excessive daytime sleepiness (total ESS score <11),
* Non-professional drivers,
* Subjects who have held their driving license for at least one year,
* Subjects affiliated to a social security scheme,
* Subjects able to understand the study,
* Subjects available to come to the 3 visits required by the study,
* Free, informed and written consent signed

Exclusion Criteria:

* Pathologies that can induce excessive daytime sleepiness: untreated narcolepsy or idiopathic hypersomnia, untreated restless legs syndrome, untreated periodic leg movement syndrome,
* Chronic insomnia disorder,
* Excessive alcohol consumption (> 2 glasses per day) during the last 6 months,
* Excessive consumption of coffee, tea or cola-type caffeinated beverages (> 5 cups/day),
* Severe pathologies involving the vital prognosis in the short term,
* Uncontrolled endocrine pathologies (dysthyroidism, diabetes),
* All progressive cardiac pathologies, treated or untreated,
* All progressive neurological conditions treated or not (brain tumor, epilepsy, migraine, stroke, sclerosis, myoclonus, chorea, neuropathy, muscular dystrophies, myotonic dystrophy, etc.),
* Substance dependence,
* Shift workers or night workers who have performed on-call or on-call duty in the last 72 hours,
* Patients taking psychotropic drugs (antidepressants, antihistamines),
* Long-term treatment with benzodiazepines and z-drugs,
* Patients on cardiotropic,
* Deprived of liberty by a judicial or administrative decision,
* Pregnant or breastfeeding woman,
* Subject under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in Objective Sleepiness Scale (OSS) during extended wakefulness | Once every 4 hours during SDP1 and SDP2 wakefulness
  OSS is based on the visual analysis of electrophysiological variables (EEG (C4, O2, C3, P3), 1 vertical EOG and 1 horizontal EOG).
  Each state of drowsiness (score) corresponds to a specific EEG activity accompanied by well-differentiated blinking and eye movements

SECONDARY OUTCOMES:
Change in Karolinska sleepiness scale (KSS) during extended wakefulness | 12 assessments every 4 hours during SDP1 and SDP2 wakefulness
  The KSS is a self-administered questionnaire that measures, on a 10 point Likert scale ranging from=1 to "fully awake" to 10 ="extremely drowsy". This measure has very good external validity on EEG synchronization measures and on the cognitive and behavioral performance of subject in relation to his or her ability to maintain wakefulness.
Change in sleep onset mesured by Maintenance of Wakefulness Test (MWT) during extended wakefulness | Once every 4 hours during SDP1 and SDP2 wakefulness
  This is test ability to stay awake in laboratory conditions conductive to falling asleep. The sleep onset latency is obtained during an electrophysiological test (EEG, EMG and EOG).
Change in number of inappropriate line crossings (driving performance) during extended wakefulness | Once every 4 hours during SDP1 and SDP2 wakefulness
  On the driving simulator the subjects will drive on a highway scenario representing a reconstruction of the real highway. Number of inappropriate line crossings (ILC) will mesured.
  An ILC was recorded when the car crossed a right or left lateral lane marker, whatever the duration and the amplitude of the crossing. Exceptions were overtaking manoeuvres or some other necessary driving action.
Change in Standard deviation of the lateral position of the car (driving performance) during extended wakefulness | Once every 4 hours during SDP1 and SDP2 wakefulness
  On the driving simulator the subjects will drive on a highway scenario representing a reconstruction of the real highway. Standard deviation of the lateral position of the car (SDLP in cm) will mesured.
  Lateral Position was defined as being 0 when the car was in the center of the lane, with positive value to the right and negative values to the left.
Change Sustained and selective attention during extended wakefulness | Once every 4 hours during SDP1 and SDP2 wakefulness
  The reaction time of subject to the presentation of a "target" stimulus (Continuous Performance Test, CPT)
Change in Vigilance during extended wakefulness | Once every 4 hours during SDP1 and SDP2 wakefulness
  The test examines the ability to concentrate and maintain attention over a long period (30mn) (TAP vigilance test)
Change in Simple reaction time test (PVT) during extended wakefulness | 1 time every 4 hours during SDP1 and SDP2 wakefulness
  Reaction-timed task that measures the consistency with which subjects respond to a visual stimulus.
Change in conscious experience during extended wakefulness | 5 assessments every 4 hours during SDP1 and SDP2 wakefulness
  Questionnaire suggests participant's attention and thoughts were entirely focused on task-related stimuli
Munich Chorotype Questionnaire | Once time during inclusion. Visit V0
  The Munich Chorotype Questionnaire (MCTQ) quantifies the chronotype according to the phase of entrainment based on the reported the mid-time of sleep; The MCTQ parameters are mid-sleep on weekdays (MSW in hr), mid-sleep on free days (MSF in hr) and mid-sleep on free days corrected for sleep debt on weekdays (MSFsc in hr). The MSFsc score (used as a chronotype indicator) represents a continuum of circadian preference, with an increasing tendency toward the evening type. MCTQ parameters are represented by hours, ranging from 0 hour (extreme morningness) to 12 hours (extreme eveningness).
Horne and Ostberg morning/evening questionnaire (MEQ) | Once time during inclusion. Visit V0
  The Horne and Ostberg morning/evening questionnaire (MEQ) quantifies the chronotype.
  The MEQ contains19 questions on life preferences (activity, sleep-wake cycle, meals) and the state of fatigue and drowsiness at certain times of the day. The MEQ score ranges from 16-86, with evening type ranging from16-41, neither or intermediate type from 42-58, and morning type from 59-86.
Daydreaming frequency scale | Once time during inclusion. Visit V0
  To assess participants' general tendency to daydream in daily life
Total sleep time (PSG) | 2 times before SDP1 and SDP2
  Total sleep time, the number of minutes asleep in bed after "lights off", will be calculated using a polysomnographic recording (PSG). EEG, EOG and EMG will be recorded during sleep.
Sleep onset latency (PSG) | 2 times before SDP1 and SDP2
  Sleep onset latency, the minutes from lights off to sleep onset, will be calculated using a polysomnographic recording (PSG). EEG, EOG and EMG will be recorded during sleep.
Sleep efficiency (PSG) | 2 times before SDP1 and SDP2
  Sleep efficiency, the ratio of the total time spent asleep (total sleep time) in a night compared to the total amount of time spent in bed, will be calculated using a polysomnographic recording (PSG). EEG, EOG and EMG will be recorded during sleep.
Amount of sleep stages (PSG) | 2 times before SDP1 and SDP2
  Amount of N1,N2,N3 and R stage (expressed in p% of TST) will be calculated using a polysomnographic recording (PSG). EEG, EOG and EMG will be recorded during sleep.
Wake after sleep onset (PSG) | 2 times before SDP1 and SDP2
  Wake after sleep onset, number of minutes scored as wake from sleep onset to the last minute scored as sleep while in bed, will be calculated using a polysomnographic recording (PSG). EEG, EOG and EMG will be recorded during sleep.
Total sleep time (actigraphy) | 2 times before SDP1 and SDP2
  Total sleep time, the number of minutes asleep in bed after "lights off", will be calculated using an actigraph (wearable sleep test that tracks wrist movements)
Sleep onset latency (actigraphy) | 2 times before SDP1 and SDP2
  Sleep onset latency, the minutes from lights off to sleep onset, will be calculated using an actigraph (wearable sleep test that tracks wrist movements)
Sleep efficiency (actigraphy) | 2 times before SDP1 and SDP2
  Sleep efficiency, the ratio of the total time spent asleep (total sleep time) in a night compared to the total amount of time spent in bed will be calculated using an actigraph (wearable sleep test that tracks wrist movements)
Wake after sleep onset (actigraphy) | 2 times before SDP1 and SDP2
  Wake after sleep onset, number of minutes scored as wake from sleep onset to the last minute scored as sleep while in bed will be calculated using an actigraph (wearable sleep test that tracks wrist movements)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Arthur Micoulaud-Franchi, MD/PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No